CLINICAL TRIAL: NCT02255513
Title: A Phase III Clinical Endpoint Evaluation Study Examining the Safety and Efficacy of HLD200 in Pediatric Subjects With Attention-Deficit Hyperactivity Disorder.
Brief Title: A Trial Evaluating the Efficacy and Safety of HLD200 in Children With ADHD
Acronym: CEES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ironshore Pharmaceuticals and Development, Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HLD200-106
Record Dates: First submitted 2014-05-29; First posted 2014-10-02 (Estimated); Results first posted 2021-02-10 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- HLD200 (Experimental): HLD200 (methylphenidate hydrochloride) 20, 40, 60, 80, or 100 mg capsules
  Subjects were allowed to titrate to their optimal HLD200 dose during a 6 week open-label, treatment optimization phase before being randomized to continue their HLD200 treatment over an one week double-blind, placebo-controlled phase. HLD200 was administered orally, once daily each evening.
  Interventions: Drug: HLD200
- Placebo (Placebo Comparator): Placebo capsules (dose matched to HLD200 capsules)
  Subjects were allowed to titrate to their optimal HLD200 dose during a 6 week open-label, treatment optimization phase before being randomized to receive placebo treatment over a one week double-blind, placebo-controlled phase. Treatments were administered orally, once daily each evening.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HLD200
  Other Names: methylphenidate hydrochloride (MPH)
  Arms: HLD200
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will examine the efficacy and safety of HLD200 in patients age 6-12 years with ADHD using a classroom study design.

DETAILED DESCRIPTION:
The study consists of two distinct treatment phases. The first is the 6-week open-label, treatment optimization phase during which subjects are titrated to an optimal daily dose of HLD200. Subjects are then randomized to receive either optimal HLD200 or matched placebo treatment for an additional week prior to final testing during a laboratory school day.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children (6-12 years at study entry)
* Previous diagnosis of ADHD and confirmation using the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID)
* Able to swallow treatment capsules
* Available for entire study period
* Provision of informed consent (from the parent[s] and/or legal representative[s]) and assent (from the subject)
* Female subjects of childbearing potential (i.e., post-menarche) required to have a negative result on urine pregnancy test (and will be given specific instructions for avoiding pregnancy during trial).

Exclusion Criteria:

* Any known history or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, ophthalmologic disease
* Presence of any significant physical or organ abnormality
* Any illness during the 4 weeks before this study
* Comorbid psychiatric diagnosis that may affect subject safety or confound results (e.g., psychosis, bipolar disorder)
* Known history of severe asthma (in the opinion of the investigator) unless deemed currently controlled
* Known history of severe allergic reaction to MPH
* Known history of seizures (except febrile seizures prior to age 5), anorexia nervosa, bulimia or current diagnosis or family history of Tourette's disorder
* Subject who are severely underweight or overweight (in the opinion of the Investigator)
* Any clinical laboratory value outside of the acceptable ranges, unless deemed NCS significant per the Investigator
* Positive history for hepatitis B, hepatitis C or Human Immunodeficiency Virus (HIV)
* Positive screening for illicit drug use, and/or current health conditions or use of medications that might confound the results of the study or increase risk to the subject
* Use of prescription medications (except ADHD medications) within 7 days and over-the-counter medications (except birth control) within the 3 days preceding study enrollment, unless deemed acceptable by the Investigator and Clinical or Medical Monitor
* Participation in clinical trial with an investigational drug within the 30 days preceding study enrollment
* Current suicidal ideation or history of suicidality determined as a significant finding on the C-SSRS by the investigator (Baseline C-SSRS for adolescents; Pediatric Baseline C-SSRS for children).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2014-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ann Childress, M.D., Principal Investigator — Center for Psychiatry And Behavioral Medicine Inc.
Locations (4):
- United States (4):
  - AVIDA, Inc., Newport Beach, California
  - South Shore Psychiatric Services, PC, Marshfield, Massachusetts
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Open-label, Treatment Optimization
Arm/Group | HLD200 | Placebo
Started | 43 | 0
Completed | 43 | 0
Not Completed | 0 | 0
Period: Double Blind, Placebo-controlled
Arm/Group | HLD200 | Placebo
Started | 22 | 21
Completed | 22 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- HLD200: Double-blind, optimal dose of HLD200 for 7 days
- Placebo: Double-blind, placebo for 7 days
- Total: Total of all reporting groups
Arm/Group | HLD200 | Placebo | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 21 | 43
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.8 (1.72) | 9.5 (1.81) | 9.7 (1.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 11 | 12 | 23
Region of Enrollment [Number; unit: participants]
  United States | 22 | 21 | 43

OUTCOME MEASURES:

1. Primary Outcome: SKAMP
Description: Swanson, Kotkin, Agler, M-Flynn and Pelham (SKAMP) Combined Scores - Average of 8:00 am to 4:00 pm assessments from the laboratory school day.
  The SKAMP is a validated, 13-item, observer-rated scale designed to assess the level of impairment of classroom-observed behaviors (Wigal and Wigal, 2006). Items 1 through 4 assess subject attention; items 5 through 8 assess deportment; items 9 through 11 assess quality of work; while items 12 and 13 assess subject compliance with teacher/classroom rules. Each individual item is rated on a 7-point scale from 0 (normal, no impairment) to 6 (maximal impairment). When all individual item scores are summed together, they produce a 13-item combined score that ranges from 0 to 78, with higher scores signifying greater impairment. In the present study, the SKAMP rating scale was utilized across 6 sessions occurring at 8:00 am, 9:00 am, 10:00 am, 12:00 pm, 2:00 pm, 4:00 pm of the laboratory school day.
Time Frame: 8-hours from 8:00 am to 4:00 pm
Measure: Least Squares Mean (Standard Deviation); unit: SKAMP Combined Score
Arm/Group | HLD200 | Placebo
Number analyzed (Participants) | 22 | 21
SKAMP Combined Score | 11.8 (1.63) | 18.9 (1.67)

ADVERSE EVENTS:
Time Frame: 1 Week (Double-blind Phase)
Arm/Group | HLD200 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 7/22 | 7/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HLD200 (N=22) | Placebo (N=21)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Emotional disorder (Psychiatric disorders) | 0 (0) | 1 (2)
Initial insomnia (Psychiatric disorders) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes